CLINICAL TRIAL: NCT01969071
Title: The Effects of Levosimendan on Renal Function in Patients With Low Ejection Fraction Undergoing Mitral Valve Surgery.
Brief Title: The Effects of Levosimendan During Mitral Valve Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Baysal, MD, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: No: 2013.2/1
Record Dates: First submitted 2013-05-24; First posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-09

CONDITIONS: Mitral Valve Stenosis With Incompetence or Regurgitation
Keywords: levosimendan; mitral valve surgery; cardiopulmonary bypass; serum creatinine; estimated glomerular filtration rate; ejection fraction
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Simendan; Dobutamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levosimendan, inotropic agent (Active Comparator): In the levosimendan group, levosimendan will be used in addition to standard inotropic therapy (one or more agent including; dopamine, dobutamine, noradrenaline, adrenaline)for 24 hours.Levosimendan dosage; a loading dose of levosimendan (6 μg kg-1) will be administered after removal of the aortic cross-clamp, followed by an infusion of levosimendan at a dose of 0.1 μg kg-1 min-1.
  Interventions: Drug: Levosimendan
- Control (Active Comparator): In the control group, only standard inotropic therapy (one or more agent including; dopamine, dobutamine, noradrenaline, adrenaline)will be administered
  Interventions: Drug: Dobutamine

INTERVENTIONS:
Drug: Levosimendan — The effects of levosimendan on renal function
  Other Names: Symdax
  Arms: Levosimendan, inotropic agent
Drug: Dobutamine — Standard Inotropic agent
  Other Names: Dobutrex
  Arms: Control

SUMMARY:
The effects of levosimendan on renal function in patients with low ejection fraction undergoing mitral valve surgery will be investigated in a prospective, double-blinded, randomized clinical trial using serum creatinine (sCr)milligram in deciliter (mg/dL) values, calculated estimated glomerular filtration(eGFR)(ml/min/1.73 m2) rates and perioperative clinical follow-up parameters.

DETAILED DESCRIPTION:
Introduction:

The coronary and peripheral vasodilatory properties of levosimendan has recently been investigated in patients with heart failure. It is considered as a promising alternative to conventional inotropic agents for patients with low LVEF. However, the effects of levosimendan on renal functions in patients undergoing open heart surgeries with CPB are not well studied in randomized clinical trials.

The primary goal of our study was to investigate the effects of levosimendan on 1- renal function by evaluation of serum creatinine (mg/dL) values and calculated estimated glomerular filtration(eGFR)(ml/min/1.73 m2) rates.

Our secondary goal was to determine clinical outcomes including;

1-need for renal replacement therapy (RRT) in patients with low ejection fraction undergoing mitral valve repair or replacement surgery with cardiopulmonary bypass (CPB).

Inclusion and exclusion criterions include as listed below. Patients included into the study had a diagnosis of mitral valve insufficiency with or without coronary artery disease and a left ventricular ejection fraction (LVEF) of ≤ 45 %.

Exclusion criteria were unstable angina, diabetes mellitus treated with insulin, clinical findings of acute or chronic renal failure (serum creatinine (sCr)> 1.5 mg/dL), severe hepatic disease (alanine aminotransferase or aspartate aminotransferase > 100 U litre/L), severe chronic obstructive pulmonary disease (forced expired volume in 1 s < 50 % of predicted or < 2.0 litre), a history of prior coronary artery bypass graft (CABG) surgery or myocardial infarction (MI) within the previous month, emergent operations, patients on inotropic support before operation, aortic valvular disease, and infective endocarditis.

The study protocol:

The patients will be randomized into two groups. Randomization into two groups was performed using sealed envelopes and the sequentially numbered assignments of the participant which will be concealed in an envelope and will be opened after anesthesia induction by a health care personnel. The observers will be blinded to the inotropic protocol. Caregivers will not be blinded, but they will not participate in data collection or data interpretation.

In the levosimendan group, a loading it of levosimendan (6 μg/kg) will be administered after removal of the aortic cross-clamp, followed by an infusion of levosimendan at a dose of 0.1 μg/kg/min in addition to standard inotropic therapy (one or more agent including; dobutamine, epinephrine or norepinephrine)for 24 hours. In the control group, only standard inotropic therapy will be administered.

The need for renal replacement therapy (RRT)will be provided to all patients under the following criterions: 1- when urine output was less than 100 mL within the last 8 hours, 2- with no response to 50 mg intravenous dose of furosemide, 3- urine sodium concentration should be > 40 milliequivalent/liter (mEq/L) before administration of furosemide, 4- blood urea nitrogen (BUN) level > 50 mg/dl 5-additional presence of one or more of the following factors such as; a- increase in serum creatinine level > 50% from preoperative value, b- presence of metabolic acidosis, c- presence of hypervolemia, d- presence of hyperkalemia (potassium ion level > 5 Meq/L).

The study parameters:

The demographic data includes; age, weight, height, body mass index and gender. The cardiovascular risk factors including; diabetes mellitus, hypertension, hypercholesterolemia, obesity, history of smoking as well as history of chronic obstructive pulmonary disease and peripheral vascular disease were sought.

Echocardiographic data were performed to evaluate the ejection fraction and valvular functions by the same cardiologist using a Vivid 3 echocardiography device (Healthcare General Electronics,Hamburg,Germany) before operation and on first hour, 12 and 24 hour after operation.

Pulmonary hypertension (PH) is defined by a mean pulmonary artery pressure (MPAP) >25 mmHg at rest. The diagnosis of PH depends on direct measurement of the mean PAP by right heart catheterization. However, we used Doppler echocardiographic study to provide an estimate of the pulmonary artery systolic pressure (PASP)and mean PAP is calculated with the formula: mean PAP = 0.65 PASP + 0.55 mmHg.

The risk of operation will be evaluated using the European System for the Cardiac Operation Risk Evaluation scale (EuroSCORE).

Acute kidney injury (AKI) is defined as increase in serum creatinine from baseline by > 50 % within 48 hours postoperatively.

SCr levels will be collected on preoperative and postoperative days 1, 3 and 10 and and eGFR will be calculated according to the abbreviated Modification of Diet in Renal Disease (MDRD) equation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mitral valve insufficiency with or without coronary artery disease and a LVEF of ≤ 45 %.

Exclusion criteria:

* unstable angina,
* diabetes mellitus treated with insulin, clinical findings of acute or chronic renal failure (sCr > 1.5 mg dL-1),
* severe hepatic disease (alanine aminotransferase or aspartate aminotransferase > 100 U litre L-1),
* severe chronic obstructive pulmonary disease (forced expired volume in 1 s < 50 % of predicted or < 2.0 litre),
* a history of prior CABG surgery or myocardial infarction (MI) within the previous month,
* emergent operations,
* patients on inotropic support before operation,
* aortic valvular disease, and
* infective endocarditis.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-07; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The effects of levosimendan on renal function in patients with low ejection fraction undergoing mitral valve surgery. | Between the time period of July 1, 2009 to January 30, 2013 participants will be followed for the duration of hospital stay, an expected average of 10 days.
  The effects of levosimendan on postoperative renal function measured by serum creatinine (sCr) levels and estimated glomerular filtration rate (eGFR).

SECONDARY OUTCOMES:
The effects of levosimendan on renal function in patients with low ejection fraction undergoing mitral valve surgery. | Between the time period of July 1, 2009 to January 30, 2013 participants will be followed for the duration of hospital stay, an expected average of 10 days.
  Secondary end points were the effects of levosimendan on clinical outcomes which include the pre- and perioperative prognostic risk factors such as; 1-aortic cross-clamp time, 2- cardiopulmonary bypass time, 3- the use of inotropic support, 4-intra-aortic balloon pump, 5- prolonged mechanical ventilation, 6-development of pneumonia, 7- Perioperative myocardial infarction, 8- cerebrovascular event (stroke, transient ischemic attack), 9- atrial fibrillation and other rhythm disturbances, 10- need for renal replacement therapy (RRT), 11-reoperation secondary to bleeding, 12-intensive care unit stay and 13- hospital stay.

OTHER OUTCOMES:
The effects of levosimendan on renal function in patients with low ejection fraction undergoing mitral valve surgery | Between the time period of July 1, 2009 to January 30, 2013 all patients will be evaluated participants will be followed for the duration of hospital stay, an expected average of 10 days.
  Hemodynamic measurements include;
  1- Cardiac output, 2-cardiac index (CI), 3-mean arterial pressure (MAP), 4-heart rate (HR), were recorded just before the start of surgery, at the end of CPB, on admission to the ICU, and postoperatively at 6 and 24 h later in the ICU. Hemodynamic targets were as follows: MAP ≥70 mmHg, CI ≥ 2.0 L/min/m2 without signs of poor peripheral perfusion (oliguria, acidosis).

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Baysal, MD, Principal Investigator — Kartal Kosuyolu High Speciality Training and Research H
Locations (1):
- Kartal Kosuyolu High Speciality Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Nieminen MS, Akkila J, Hasenfuss G, Kleber FX, Lehtonen LA, Mitrovic V, Nyquist O, Remme WJ. Hemodynamic and neurohumoral effects of continuous infusion of levosimendan in patients with congestive heart failure. J Am Coll Cardiol. 2000 Nov 15;36(6):1903-12. doi: 10.1016/s0735-1097(00)00961-x. PMID 11092663
- [Background] Garcia Gonzalez MJ, Dominguez Rodriguez A. Pharmacologic treatment of heart failure due to ventricular dysfunction by myocardial stunning: potential role of levosimendan. Am J Cardiovasc Drugs. 2006;6(2):69-75. doi: 10.2165/00129784-200606020-00001. PMID 16555860
- [Background] Yilmaz MB, Yalta K, Yontar C, Karadas F, Erdem A, Turgut OO, Yilmaz A, Tandogan I. Levosimendan improves renal function in patients with acute decompensated heart failure: comparison with dobutamine. Cardiovasc Drugs Ther. 2007 Dec;21(6):431-5. doi: 10.1007/s10557-007-6066-7. Epub 2007 Oct 20. PMID 17952581
- [Result] De Hert SG, Lorsomradee S, Cromheecke S, Van der Linden PJ. The effects of levosimendan in cardiac surgery patients with poor left ventricular function. Anesth Analg. 2007 Apr;104(4):766-73. doi: 10.1213/01.ane.0000256863.92050.d3. PMID 17377079
- [Result] Hernandez A, Miranda A, Parada A. [Levosimendan reduces mortality in cardiac surgery: a systematic review and meta-analysis]. Rev Esp Anestesiol Reanim. 2012 Jan;59(1):6-11. doi: 10.1016/j.redar.2012.02.001. Epub 2012 Mar 14. Spanish. PMID 22429630
- [Result] Severi L, Lappa A, Landoni G, Di Pirro L, Luzzi SJ, Caravetta P, Cipullo P, Menichetti A. Levosimendan versus intra-aortic balloon pump in high-risk cardiac surgery patients. J Cardiothorac Vasc Anesth. 2011 Aug;25(4):632-6. doi: 10.1053/j.jvca.2011.03.001. Epub 2011 May 4. PMID 21546269
- [Result] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Result] Metra M, Nodari S, Parrinello G, Bordonali T, Bugatti S, Danesi R, Fontanella B, Lombardi C, Milani P, Verzura G, Cotter G, Dittrich H, Massie BM, Dei Cas L. Worsening renal function in patients hospitalised for acute heart failure: clinical implications and prognostic significance. Eur J Heart Fail. 2008 Feb;10(2):188-95. doi: 10.1016/j.ejheart.2008.01.011. PMID 18279773
- [Result] Haase-Fielitz A, Bellomo R, Devarajan P, Story D, Matalanis G, Dragun D, Haase M. Novel and conventional serum biomarkers predicting acute kidney injury in adult cardiac surgery--a prospective cohort study. Crit Care Med. 2009 Feb;37(2):553-60. doi: 10.1097/CCM.0b013e318195846e. PMID 19114878
- [Result] Elahi MM, Lim MY, Joseph RN, Dhannapuneni RR, Spyt TJ. Early hemofiltration improves survival in post-cardiotomy patients with acute renal failure. Eur J Cardiothorac Surg. 2004 Nov;26(5):1027-31. doi: 10.1016/j.ejcts.2004.07.039. PMID 15519198